CLINICAL TRIAL: NCT05475626
Title: Treatment Of Symptomatic Pes Planus By Sinus Tarsi Screw Versus Conical Subtalar Screw Arthroereisis- A Randomised Controlled Study
Brief Title: Treatment Of Symptomatic Pes Planus By Sinus Tarsi Screw Versus Conical Subtalar Screw Arthroereisis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Ali Hassan Abdelhamid (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Ali Hassan Abdelhamid, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Randomized controlled study
Record Dates: First submitted 2022-07-20; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Symptomatic Flexible Flat Feet

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Of Symptomatic Pes Planus By Sinus Tarsi Screw: Treatment Of Symptomatic Pes Planus
  Interventions: Procedure: Arthroereisis-

INTERVENTIONS:
Procedure: Arthroereisis- — Surgical options include soft tissue procedures, realignment osteotomies and non-fusion motion-limiting techniques.

SUMMARY:
compare the outcome of surgical treatment planus by sinus tarsi screw versus conical subtalar screw arthroereisis

DETAILED DESCRIPTION:
Pes planus occurs as a result of loss of the medial longitudinal arch, abduction of the forefoot and excessive subtalar eversion. It can broadly be categorized as rigid or flexible.(1) Flexible pes planus has no single identifiable cause and is often asymptomatic.(1-3) Patients with pesplanus had a very tight achilles tendon due to compensatory motion.(4) It can become painful and may require orthopaedic or pediatric intervention. Common treatment modalities include rest, physiotherapy, orthotics and anti-inflammatories.(1,3,5-6) Surgery is uncommon unless pain persists in spite of nonsurgical management.(5-6) Surgical options include soft tissue procedures, realignment osteotomies and non-fusion motion-limiting techniques.(1,2,6-9) Fusion of selected joints in the foot is not recommended in paediatric patients unless associated with a neuromuscular pathology.(1,5) Subtalar arthroereisis is a recognized non-fusion surgical treatment for symptomatic paediatric flexible pes planus. Arthroereisis (also arthroreisis, arthrorhisis or arthrorisis) derives from Greek, translated as to prop up or support a joint.(10) When Flexible pes planus becomes symptomatic, affecting gait and limiting quality of life, and conservative treatment such as weight reduction, physiotherapy or insoles fail, operative treatment can be considered .(7) There are two techniques for subtalar arthroereisis: (11) Insertion of an implant directly into the sinus tarsi to prevent it collapsing down. (10) Screw insertion into the lateral side of either the talus or calcaneus(12). Calcaneo-stop method with cancellous screw insertion into sinus tarsi for subtalar arthroresis is a valid procedure for this multiplanar deformity. Maintaince of correction of the deformity is achieved via a prioprioceptive mechanism. (13) The current research is the first one to compare the clinical , radiological,and patient satisfaction outcome of planovalgus cases treated with two different types of subtalar arthroereisis implants . The purpose of this prospective study is to show the best technique to achieve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

- Patients are eligible for participation in the study if

* Patients above the ages of 7years
* All patients with symptomatic pes planus
* flexible flat feet
* Not respond to conservative therapies.

Exclusion Criteria:

* Patients are excluded for participation in the study if

  * Patients were age < 7 years
  * Asymptomatic patient
  * Rigid flat feet
  * Unfit for surgery
  * Children with neuromuscular diseases, post traumatic or congenital pes planovalgus will be excluded from the study

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients above the ages of 7years
  • All patients with symptomatic pes planus
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
to identify and evaluate the comparison between two technical procedure of surgical treatment of symptomatic pes planus by sinus tarsi screw versus conical subtalar screw arthroerasis using American Orthopaedic Foot and Ankle Society scores (AOFAS) | 2 years
  American Orthopedic Foot & Ankle Society (AOFAS) ankle-hind foot score was assessed. The total AOFAS score 100 points divided to 40 points for assessment of pain, 50 points for the functional assessment " activity limitations, maximum walking distance, gait abnormality…etc" and 10 points for assessment of the alignment.

SECONDARY OUTCOMES:
): to detect the radiographic measurments change between the surgical treatment of symptomatic pes planus by sinus tarsi screw versus conical subtalar arthroerasis | 1 year
  RadiologicalEvaluation(AP&lateral)withangleevaluation:Radiographswillbe takenpreoperatively,directlypostoperatively,andatmidtermfollow-upina weight-bearingstandingposition.Thecalcanealpitch(CP)andMeary'sangle (MA;alsoreferredtoaslateraltalo-firstmetatarsalangle)willbeusedto determinefootanatomy

IPD SHARING:
Plan to Share IPD: Undecided
Treatment Of Symptomatic Pes Planus By Sinus Tarsi Screw Versus Conical Subtalar Screw Arthroereisis- A Randomised Controlled Study

REFERENCES:
- [Background] Carr JB II, Yang S, Lather LA. Pediatric pes planus: a state-of-the-art review.Pediatrics 2016;137:e20151230. 2. Dare DM, Dodwell ER. Pediatric flatfoot: cause, epidemiology, assessment, and treatment. Curr Opin Pediatr 2014;26:93-100. 3. Mosca VS. Flexible flatfoot in children and adolescents. J Child Orthop 10;4:107-121. 4. Raj MA, Tafti D, Kiel J. Pes Planus (Flat Feet). StatPearl-NCBI Bookshelf, 2020. Available from: https://www.ncbi.nlm.nih.gov/books/NBK430802/ (Accessed 29 June 2020) 5.Sheikh Taha AM, Feldman DS. Painful flexible flatfoot. Foot Ankle Clin 2015;20:693-704. 6. Bouchard M, Mosca VS. Flatfoot deformity in children and adolescents: surgical indications and management. J Am Acad Orthop Surg 2014;22:623-632. 7. Walters JL, Mendicino SS. Flexible adult flatfoot: soft tissue procedures. Clin Podiatr Med Surg 2014;31:349-355. 8. Peterson KS, Overley BD Jr, Beideman TC. Osteotomies for the flexible adult acquired flatfoot disorder. Clin Podiatr Med Surg 2015;32:389-403. 9. Abubeih ,Hossam MA.,Wael El-Adly ,and Kotb,M.M. Modified calcaneo-stop screw method for treatment of symptomatic pediatric flexible flatfoot deformity . Current Orthopaedic Practice 26.6 (2015);614-618. 10. Medical Dictionary. Arthroereisis. The Free Dictionary. https://medical-dictionary. The free dictionary .com/arthroereisis (date last accessed 5 July 2018). 11. Chambers EF. An operation for the correction of flexible flat feet of adolescents. West J Surg Obstet Gynecol 1946;54:77-86. 12. Shah NS, Needleman RL, Bokhari O, Buzas D. 2013 subtalar arthroereisis survey: the current practice patterns of members of the AOFAS. Foot Ankle Spec 2015;8: 180-185 13. Staheli L. Planovalgus foot deformity.Current status.Journal of the American Podiatric Medical Association 1999;89(2): 94-9. 14. Ritchie GW and Keim HA .A radiographic analysis of major foot deformities.Canad Med Ass J Oct 1963;Vol 91 .
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK430802